CLINICAL TRIAL: NCT03359863
Title: Pirfenidone for Restrictive Chronic Lung Allograft Dysfunction
Acronym: PIRCLAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-20710
Record Dates: First submitted 2017-11-15; First posted 2017-12-02 (Actual); Results first posted 2023-01-09 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Restrictive Chronic Lung Allograft Dysfunction; Lung Transplant Rejection
MeSH Terms: interventions — pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): Subjects will receive Pirfenidone as part of treatment for their restrictive chronic lung allograft dysfunction (RCLAD).
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Subjects will receive pirfenidone for 52 weeks, titrated to 2403 mg/day (3 capsules, 3× daily) after a 4-week titration period (1 capsule, 3x daily for 2 weeks, 2 capsules, 3x daily for 2 weeks) for a total of 56 weeks of pirfenidone. Eligible participants will continue pirfenidone beyond 56 weeks.
  Other Names: Esbriet

SUMMARY:
Despite advances in lung transplantation, the median survival remains only 55% at 5 years. The main limitation to long term survival is the development of chronic lung allograft dysfunction. In approximately 30% of cases, chronic lung allograft dysfunction has a restrictive phenotype (RCLAD) characterized by fibrosis with rapid progression to respiratory failure. Approximately 60% of patients with RCLAD die within one year, as currently there are no therapies available.

RCLAD, like Idiopathic Pulmonary Fibrosis (IPF), is characterized by fibroblast proliferation, extracellular matrix deposition, and architectural distortion leading to progressive lung scarring and death. Given their similarities, there is keen interest in the international transplant community to investigate whether the anti-fibrotic drug pirfenidone can slow the progression of RCLAD as it does of IPF. Pirfenidone has been proved to be safe and effective in patients with IPF, and is approved by the Food and Drug Administration.

This protocol will evaluate the safety and tolerability of pirfenidone in lung transplant recipients with RCLAD. Transplant recipients take carefully adjusted immunosuppressive medications for life to prevent rejection of the allograft. Current literature suggests the dose of tacrolimus, the main anti-rejection drug, may need to be adjusted when taken in combination with pirfenidone. The investigators will assess the side effects of pirfenidone in combination with the immunosuppressive regimen and determine the magnitude of the adjustment in tacrolimus dose. The results of this pilot study will provide the foundation for a multicenter randomized control trial to evaluate the efficacy of pirfenidone in slowing the progression of RCLAD.

DETAILED DESCRIPTION:
Despite advances in lung transplantation, median survival remains only 55% at 5 years. The primary cause of death is chronic lung allograft dysfunction (CLAD), occurring in 43% of recipients at 5 years. Recently, it has been recognized that CLAD can have an obstructive (BOS) or a restrictive (RCLAD) phenotype, also known as restrictive allograft syndrome (RAS), and that both may coexist. These phenotypes differ not only in their spirometric, radiographic and histologic features but also in their rates of progression and survival. Thus, there is a critical need to find therapies other than re-transplantation, which remains the only effective therapeutic option and explore the pathobiology driving RCLAD.

RCLAD shares features with Idiopathic Pulmonary Fibrosis (IPF), including its progressive and lethal course, extracellular matrix deposition, architectural distortion, fibroblast proliferation, and short telomeres in lung epithelial cells. These common features suggest RCLAD and IPF may share molecular pathogenesis. As a result, some have explored using FDA approved anti-fibrotic medications for IPF in RCLAD in case reports.

This proposal aims to gather the preliminary data needed to design a multicenter randomized controlled trial (RCT) of pirfenidone for RCLAD. To do so, the investigators first need evidence of tolerability, to understand drug interactions with the immunosuppressive regimen used to maintain allograft function and early evidence that pirfenidone may slow FVC decline and radiographic progression in RCLAD.

Evidence that pirfenidone is well tolerated in transplant recipients and that it slows the progression of RCLAD would be paradigm shifting. Further, identifying subjects at risk for RCLAD before the onset of spirometric changes would allow to start therapeutic interventions sooner, maximizing their benefit. Finding biomarkers that predict response to pirfenidone would identify patients most likely to benefit.

ELIGIBILITY:
Inclusion Criteria:

* Subject who underwent bilateral lung transplantation at University of California San Francisco (UCSF) and have a diagnosis of RCLAD based on the International Heart and Lung Transplant (ISHLT) classification. The diagnosis of RCLAD is based on spirometry (Forced Expiratory Volume in 1 second (FEV1) ≤ 80% and FVC ≤ 80% of best post-transplant baseline) and CT scan (e.g. pleuroparenchymal fibroelastosis) findings.

Exclusion Criteria:

* FVC decline related to non-RCLAD causes (e.g. pulmonary edema, pleural effusion, etc).
* Patients with any severe comorbidity complicating RCLAD which might determine their prognosis and functional level (e.g. active malignant disease) within the last 12 months
* Patients who have resumed smoking after transplantation
* Renal insufficiency (creatinine clearance < 30 ml/min calculated by the CKD-Epi formula)
* Total bilirubin above the upper limit of the normal range (ULN)
* Aspartate or alanine aminotransferase (AST or ALT) > 3 times the ULN.
* Known allergy of hypersensitivity to Pirfenidone
* Pregnancy
* Ongoing use or expected use of any of the following therapies:
* Strong inhibitors of CYP1A2 (e.g. fluvoxamine or enoxacin).
* Moderate inhibitors of CAYP1A2 (e. g. mexiletine, thiabendazole, or phenylpropanolamine). Ciprofloxacin will be allowed only at doses equal or less than 500 mg BID.
* Inability to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aida A Venado Estrada, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valapour M, Skeans MA, Smith JM, Edwards LB, Cherikh WS, Callahan ER, Israni AK, Snyder JJ, Kasiske BL. Lung. Am J Transplant. 2016 Jan;16 Suppl 2:141-68. doi: 10.1111/ajt.13671. PMID 26755267
- [Background] Verleden GM, Raghu G, Meyer KC, Glanville AR, Corris P. A new classification system for chronic lung allograft dysfunction. J Heart Lung Transplant. 2014 Feb;33(2):127-33. doi: 10.1016/j.healun.2013.10.022. Epub 2013 Oct 24. PMID 24374027
- [Background] Saito T, Horie M, Sato M, Nakajima D, Shoushtarizadeh H, Binnie M, Azad S, Hwang DM, Machuca TN, Waddell TK, Singer LG, Cypel M, Liu M, Paul NS, Keshavjee S. Low-dose computed tomography volumetry for subtyping chronic lung allograft dysfunction. J Heart Lung Transplant. 2016 Jan;35(1):59-66. doi: 10.1016/j.healun.2015.07.005. Epub 2015 Aug 13. PMID 26342441
- [Background] Pakhale SS, Hadjiliadis D, Howell DN, Palmer SM, Gutierrez C, Waddell TK, Chaparro C, Davis RD, Keshavjee S, Hutcheon MA, Singer LG. Upper lobe fibrosis: a novel manifestation of chronic allograft dysfunction in lung transplantation. J Heart Lung Transplant. 2005 Sep;24(9):1260-8. doi: 10.1016/j.healun.2004.08.026. PMID 16143243
- [Background] Ofek E, Sato M, Saito T, Wagnetz U, Roberts HC, Chaparro C, Waddell TK, Singer LG, Hutcheon MA, Keshavjee S, Hwang DM. Restrictive allograft syndrome post lung transplantation is characterized by pleuroparenchymal fibroelastosis. Mod Pathol. 2013 Mar;26(3):350-6. doi: 10.1038/modpathol.2012.171. Epub 2012 Sep 28. PMID 23018877
- [Background] Sato M, Hwang DM, Waddell TK, Singer LG, Keshavjee S. Progression pattern of restrictive allograft syndrome after lung transplantation. J Heart Lung Transplant. 2013 Jan;32(1):23-30. doi: 10.1016/j.healun.2012.09.026. PMID 23260703
- [Background] Sato M, Waddell TK, Wagnetz U, Roberts HC, Hwang DM, Haroon A, Wagnetz D, Chaparro C, Singer LG, Hutcheon MA, Keshavjee S. Restrictive allograft syndrome (RAS): a novel form of chronic lung allograft dysfunction. J Heart Lung Transplant. 2011 Jul;30(7):735-42. doi: 10.1016/j.healun.2011.01.712. Epub 2011 Mar 17. PMID 21419659
- [Background] Todd JL, Jain R, Pavlisko EN, Finlen Copeland CA, Reynolds JM, Snyder LD, Palmer SM. Impact of forced vital capacity loss on survival after the onset of chronic lung allograft dysfunction. Am J Respir Crit Care Med. 2014 Jan 15;189(2):159-66. doi: 10.1164/rccm.201306-1155OC. PMID 24325429
- [Background] Verleden SE, de Jong PA, Ruttens D, Vandermeulen E, van Raemdonck DE, Verschakelen J, Vanaudenaerde BM, Verleden GM, Vos R. Functional and computed tomographic evolution and survival of restrictive allograft syndrome after lung transplantation. J Heart Lung Transplant. 2014 Mar;33(3):270-7. doi: 10.1016/j.healun.2013.12.011. Epub 2013 Dec 17. PMID 24461432
- [Background] Verleden GM, Vos R, Verleden SE, De Wever W, De Vleeschauwer SI, Willems-Widyastuti A, Scheers H, Dupont LJ, Van Raemdonck DE, Vanaudenaerde BM. Survival determinants in lung transplant patients with chronic allograft dysfunction. Transplantation. 2011 Sep 27;92(6):703-8. doi: 10.1097/TP.0b013e31822bf790. PMID 21836537
- [Background] Woodrow JP, Shlobin OA, Barnett SD, Burton N, Nathan SD. Comparison of bronchiolitis obliterans syndrome to other forms of chronic lung allograft dysfunction after lung transplantation. J Heart Lung Transplant. 2010 Oct;29(10):1159-64. doi: 10.1016/j.healun.2010.05.012. Epub 2010 Jun 26. PMID 20580267
- [Background] Verleden SE, Ruttens D, Vandermeulen E, Bellon H, Dubbeldam A, De Wever W, Dupont LJ, Van Raemdonck DE, Vanaudenaerde BM, Verleden GM, Benden C, Vos R. Predictors of survival in restrictive chronic lung allograft dysfunction after lung transplantation. J Heart Lung Transplant. 2016 Sep;35(9):1078-84. doi: 10.1016/j.healun.2016.03.022. Epub 2016 Apr 16. PMID 27212563
- [Background] Verleden SE, Todd JL, Sato M, Palmer SM, Martinu T, Pavlisko EN, Vos R, Neyrinck A, Van Raemdonck D, Saito T, Oishi H, Keshavjee S, Greer M, Warnecke G, Gottlieb J, Haverich A. Impact of CLAD Phenotype on Survival After Lung Retransplantation: A Multicenter Study. Am J Transplant. 2015 Aug;15(8):2223-30. doi: 10.1111/ajt.13281. Epub 2015 Apr 30. PMID 25940517
- [Background] Fernandez IE, Heinzelmann K, Verleden S, Eickelberg O. Characteristic patterns in the fibrotic lung. Comparing idiopathic pulmonary fibrosis with chronic lung allograft dysfunction. Ann Am Thorac Soc. 2015 Mar;12 Suppl 1:S34-41. doi: 10.1513/AnnalsATS.201410-476MG. PMID 25830833
- [Background] Alder JK, Chen JJ, Lancaster L, Danoff S, Su SC, Cogan JD, Vulto I, Xie M, Qi X, Tuder RM, Phillips JA 3rd, Lansdorp PM, Loyd JE, Armanios MY. Short telomeres are a risk factor for idiopathic pulmonary fibrosis. Proc Natl Acad Sci U S A. 2008 Sep 2;105(35):13051-6. doi: 10.1073/pnas.0804280105. Epub 2008 Aug 27. PMID 18753630
- [Background] Vos R, Verleden SE, Ruttens D, Vandermeulen E, Yserbyt J, Dupont LJ, Van Raemdonck DE, De Raedt N, Gheysens O, De Jong PA, Verleden GM, Vanaudenaerde BM. Pirfenidone: a potential new therapy for restrictive allograft syndrome? Am J Transplant. 2013 Nov;13(11):3035-40. doi: 10.1111/ajt.12474. Epub 2013 Sep 18. PMID 24102752
- [Background] Suhling H, Bollmann B, Gottlieb J. Nintedanib in restrictive chronic lung allograft dysfunction after lung transplantation. J Heart Lung Transplant. 2016 Jul;35(7):939-40. doi: 10.1016/j.healun.2016.01.1220. Epub 2016 Feb 9. No abstract available. PMID 26996931
- [Background] Lancaster L, Albera C, Bradford WZ, Costabel U, du Bois RM, Fagan EA, Fishman RS, Glaspole I, Glassberg MK, King TE Jr, Lederer DJ, Lin Z, Nathan SD, Pereira CA, Swigris JJ, Valeyre D, Noble PW. Safety of pirfenidone in patients with idiopathic pulmonary fibrosis: integrated analysis of cumulative data from 5 clinical trials. BMJ Open Respir Res. 2016 Jan 12;3(1):e000105. doi: 10.1136/bmjresp-2015-000105. eCollection 2016. PMID 26835133
- [Background] Khanna D, Albera C, Fischer A, Khalidi N, Raghu G, Chung L, Chen D, Schiopu E, Tagliaferri M, Seibold JR, Gorina E. An Open-label, Phase II Study of the Safety and Tolerability of Pirfenidone in Patients with Scleroderma-associated Interstitial Lung Disease: the LOTUSS Trial. J Rheumatol. 2016 Sep;43(9):1672-9. doi: 10.3899/jrheum.151322. Epub 2016 Jul 1. PMID 27370878
- [Background] King TE Jr, Bradford WZ, Castro-Bernardini S, Fagan EA, Glaspole I, Glassberg MK, Gorina E, Hopkins PM, Kardatzke D, Lancaster L, Lederer DJ, Nathan SD, Pereira CA, Sahn SA, Sussman R, Swigris JJ, Noble PW; ASCEND Study Group. A phase 3 trial of pirfenidone in patients with idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2083-92. doi: 10.1056/NEJMoa1402582. Epub 2014 May 18. PMID 24836312

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 10
Completed | 5
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Pirfenidone
Description: The primary outcome will be the number of subjects that discontinue pirfenidone due to a treatment emergent adverse event (TEAE)
Time Frame: From initiation of pirfenidone until discontinuation or until 56 weeks, which ever comes first.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
Participants | 3

2. Primary Outcome: Conversion Ratio of Tacrolimus Dose
Description: The outcome will be the ratio of tacrolimus-while-taking-pirfenidone to tacrolimus-before-pirfenidone corrected for the subject's specific steady-state tacrolimus concentration.
Time Frame: From initiation of pirfenidone until discontinuation or until 56 weeks, which ever comes first.
Measure: Mean (Standard Deviation); unit: conversion ratio
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
conversion ratio | 1.1 (0.6)

3. Secondary Outcome: Annual Change in Forced Vital Capacity (FVC)
Description: The investigators will evaluate change in FVC from baseline to 1 year after pirfenidone start based on pulmonary function tests done as part of routine clinical care (usually obtained every 3 months) or death, whichever comes first.
Time Frame: FVC change from baseline (screening) to 1 year or death, whichever comes first.
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
mL | -63.3 [-245.5 to 118.9]

4. Secondary Outcome: Annual Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: The investigators will evaluate change in FEV1 from baseline to 1 year based on pulmonary function tests done as part of routine clinical care (usually obtained every 3 months) or death, whichever comes first.
Time Frame: FEV1 change from baseline (screening) to 1 year or death, whichever comes first.
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
mL | -87.8 [-237.3 to 61.8]

5. Secondary Outcome: Annual Change in Percent of Lung Affected by Reticulation on Chest CT Scan
Description: The investigators will evaluate the annual change in percent of lung affected by reticulation comparing the chest CT scan at screening and a 1-year follow up CT scan performed as part of routine clinical care or death, whichever comes first.
Time Frame: Change between chest CT at screening and in 1-year follow up CT scan performed as part of routine clinical care or death, whichever comes first.
Measure: Mean (95% Confidence Interval); unit: percentage of lung affected
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
percentage of lung affected | 3 [-0.8 to 6.8]

6. Secondary Outcome: Annual Change in Traction Bronchiectasis Score on Chest CT Scan
Description: The investigators will evaluate the change in traction bronchiectasis score on chest CT scan at screening and in a 1-year follow up CT scan performed as part of routine clinical care or death, whichever comes first. The extent of traction bronchiectasis was first scored in each of the six lung lobes separately (right upper, middle, and lower lobes, and left upper, lingula, and lower lobes) as 0-absent, 1-mild, 2-moderate, or 3-severe, and then summed into a total traction bronchiectasis score [range 0-18 points], with higher values reflecting greater extent of traction bronchiectasis.
Time Frame: Change between Chest CT at screening and 1-year follow up CT scan performed as part of routine clinical care or death, whichever comes first.
Measure: Mean (95% Confidence Interval); unit: points
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
points | 0.8 [-0.1 to 1.7]

ADVERSE EVENTS:
Time Frame: Up to 56 weeks for each participant
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 3/10
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=10)
Hospitalization for COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1
Hospitalization for neck pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness and Vomiting (Gastrointestinal disorders) | 1
Hospitalization for pseudomonas pneumonia, CMV viremia and epigastric pain (Gastrointestinal disorders) | 1
Hospitalization for cellulitis of the neck (Skin and subcutaneous tissue disorders) | 2
Hospitalization for progressive respiratory failure leading to retransplant (Respiratory, thoracic and mediastinal disorders) | 2
Hospitalization for herpes zoster ophtalmicus (Eye disorders) | 1
Hospitalization for pneumonia with Aspergillus (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=10)
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Diarrhea (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 9
Dizziness/Lightheadedness (General disorders) | 6
Neuropathy - sensory (Nervous system disorders) | 4
Headache (General disorders) | 8
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Inner ear / hearing (Ear and labyrinth disorders) | 4
Photosensitivity / Phototoxicity (Skin and subcutaneous tissue disorders) | 2
Neuropathy - motor (Nervous system disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Alopecia (General disorders) | 5
Hypertension (Cardiac disorders) | 9
Mood alteration (Psychiatric disorders) | 6
Ocular / visual (Eye disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 3
Wound - infections (Infections and infestations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Confusion (Nervous system disorders) | 2
Fever (Infections and infestations) | 1
Rash / desquamation (Skin and subcutaneous tissue disorders) | 1
Neuropathy - cerebellar (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Small, single-center cohort with an open-label intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/63/NCT03359863/Prot_SAP_002.pdf